CLINICAL TRIAL: NCT05414708
Title: Art Therapy and Emotional Well Being in Military Populations With Posttraumatic Stress Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13476
Record Dates: First submitted 2021-12-15; First posted 2022-06-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-08

CONDITIONS: PTSD; Military Activity; Post-Traumatic Headache; Posttraumatic Stress Disorder; Posttraumatic Stress Disorder, Delayed Onset; Sleep Disturbance; Nightmare; Irritable Mood; Anger; Combat and Operational Stress Reaction; Combat Stress Disorders; Military Family; Military Operations; Emotional Regulation; Emotion Processing
Keywords: PTSD; Military; Art Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Post-Traumatic Headache; Parasomnias; Combat Disorders; Emotional Regulation | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Art Therapy Arm (Experimental): 8 weeks of individual art therapy
  Interventions: Behavioral: Art Therapy

INTERVENTIONS:
Behavioral: Art Therapy — During the art research intervention session, the art therapist will walk you through the creation of various types of art and may spend time asking you about the artwork, how you are felling, as well as your past experiences.

SUMMARY:
Art therapy is used across the Military Health System for treatment of posttraumatic symptoms, but there is limited research on how art therapy is able to restore emotional expression and regulation in service members. This research hopes to learn about the effects of art therapy on emotional expression and regulation in service members as well as the neurological systems at work. If a participant chooses to be in this study, he or she will attend eleven sessions over a period of six to eight months. The first session will be an interview and self-assessment questionnaires to collect information on a variety of symptoms, experiences, and personality traits, and an MRI scan. During the MRI scan, participants will be asked to perform a task where they will be shown a series of neutral and negative images. The following eight sessions will be one-hour art therapy sessions with a certified art therapist. The tenth session will consist of the same self-assessment questionnaires and another MRI scan. The final session will consist of some of the same questionnaires from the tenth visit, as well as a qualitative interview done virtually three months after the tenth visit.

DETAILED DESCRIPTION:
Art Therapy is used across the Military Health System (MHS) as part of interdisciplinary treatment programs with great success, but there is limited research on how this art therapy works. Therefore, the purpose of this research is to learn about the effects of art therapy on emotional expression and regulation in service members as well as the impact of art therapy on brain systems. If a participant chooses to be in this study he or she will attend eleven sessions over a period of six to eight months. The first session and tenth sessions of this research study will include interviews and self-assessment questionnaires to collect information on a variety of symptoms, experiences, and personality traits, and a magnetic resonance imaging (MRI) scan. During the MRI scan, participants will be asked to perform a task where they will be shown a series of neutral and negative images. These sessions will be about 2.5 to 3 hours. The sessions two through nine will include a one-hour art therapy sessions with a certified art therapist. The art therapy sessions are also considered research interventions. The eleventh and final session will consist of some of the same questionnaires from the tenth visit, as well as a qualitative interview done virtually three months after the tenth visit.

There is the risk that participants may experience increased psychological or emotional distress or frustration when discussing traumatic events during either the art research intervention sessions or during the questionnaires or interviews. Participants may experience a reduction in symptoms associated with posttraumatic stress (PTS), mild traumatic brain injury (mTBI), and/or other psychological heath disorders through the art therapy process. However, there is no guarantee that participants will benefit from being in this research. As an alternative to this research, participants can talk to your physician about art therapy or other therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* DEERS Eligible
* Active Duty or Veteran separated within the past 10 years
* Significant posttraumatic stress symptoms (score of >/=31 on the PCL-5)

Exclusion Criteria:

* History of moderate, severe, or penetrating brain injury
* History of psychotic disorder, bipolar disorder, or active suicidal or homicidal ideation
* History of multiple sclerosis, Huntington's disease, or Alzheimer's disease
* History of stroke or myocardial infarction
* History of brain tumor
* History of seizures
* Contradictions for MRI (for example, participants will be excluded for pregnancy, metal implants or suspected shrapnel, aneurysm/intracranial clips, cardiac pacemakers or implanted programmable devices or pumps)
* Unable to provide informed consent
* History of previous exposure to art therapy
* Active substance use disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Primary Outcome Measure is analysis of functional neuroimaging metrics | Baseline
  The primary outcome measure is the analysis of resting state and task based functional MRI data which include but functional connectivity measures between brain regions at rest and during the task as well as functional activation patterns during the task.
  MRI and a series of task based fMRI sequences.
The Primary Outcome Measure is analysis of functional neuroimaging metrics | Through study completion, an average of 14 weeks
  The primary outcome measure is the analysis of resting state and task based functional MRI data which include but functional connectivity measures between brain regions at rest and during the task as well as functional activation patterns during the task.
  MRI and a series of task based fMRI sequences.

SECONDARY OUTCOMES:
Toronto Alexithymia Scale (TAS-20) | Baseline
  A 20-item instrument that measures alexithymia defined as trouble identifying and describing emotions. A 20-item instrument that measures alexithymia defined as trouble identifying and describing emotions. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree.
Toronto Alexithymia Scale (TAS-20) | Through study completion, an average of 14 weeks
  A 20-item instrument that measures alexithymia defined as trouble identifying and describing emotions. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree.
PTSD Checklist for the Diagnostics and Statistics Manual Five (DSM-V) (PCL-5) | Baseline
  A 20-item self-report measure of the 20 DSM-5 symptoms of PTSD. Respondents rate how much they were "bothered by that problem in the past month". Items are rated on a scale ranging from 0 ("not at all") to 4 ("extremely")
PTSD Checklist for the Diagnostics and Statistics Manual Five (DSM-V) (PCL-5) | Through study completion, an average of 14 weeks
  A 20-item self-report measure of the 20 DSM-5 symptoms of PTSD. Respondents rate how much they were "bothered by that problem in the past month". Items are rated on a scale ranging from 0 ("not at all") to 4 ("extremely")
PTSD Checklist for the Diagnostics and Statistics Manual Five (DSM-V) (PCL-5) | Study completion, an average of six to eight months
  A 20-item self-report measure of the 20 DSM-5 symptoms of PTSD. Respondents rate how much they were "bothered by that problem in the past month". Items are rated on a scale ranging from 0 ("not at all") to 4 ("extremely")
Neurobehavioral Symptoms Inventory (NSI) | Baseline
  A self-reported questionnaire that measures common post concussive symptoms. The severity of each symptom as experienced in the last two weeks is rated on a scale (0) none to (4) very severe
Neurobehavioral Symptoms Inventory (NSI) | Through study completion, an average of 14 weeks
  A self-reported questionnaire that measures common post concussive symptoms. The severity of each symptom as experienced in the last two weeks is rated on a scale (0) none to (4) very severe
Neurobehavioral Symptoms Inventory (NSI) | Study completion, an average of six to eight months
  A self-reported questionnaire that measures common post concussive symptoms. The severity of each symptom as experienced in the last two weeks is rated on a scale (0) none to (4) very severe
General Self Efficacy Scale (GSES) | Baseline
  A self-report questionnaire that predicts coping with and adapting to stressful life event. The extent to which the participant agrees with each statement is measured on a scale of 1 (not true at all) to 4 (exactly true).
General Self Efficacy Scale (GSES) | Through study completion, an average of 14 weeks
  A self-report questionnaire that predicts coping with and adapting to stressful life event. The extent to which the participant agrees with each statement is measured on a scale of 1 (not true at all) to 4 (exactly true).
General Self Efficacy Scale (GSES) | Study completion, an average of six to eight months
  A self-report questionnaire that predicts coping with and adapting to stressful life event. The extent to which the participant agrees with each statement is measured on a scale of 1 (not true at all) to 4 (exactly true).
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  A self-rated questionnaire that screens for generalized anxiety disorder. A recommended threshold for further evaluation is a score of 10 or greater
Generalized Anxiety Disorder-7 (GAD-7) | Through study completion, an average of 14 weeks
  A self-rated questionnaire that screens for generalized anxiety disorder. A recommended threshold for further evaluation is a score of 10 or greater
Generalized Anxiety Disorder-7 (GAD-7) | Study completion, an average of six to eight months
  A self-rated questionnaire that screens for generalized anxiety disorder. A recommended threshold for further evaluation is a score of 10 or greater
Self-Regulation Questionnaire (SRQ) | Baseline
  A self-report questionnaire that measures the ability to develop, implement, and flexibly maintain planned behavior. The extent to which the participant agrees with each statement is rated on a scale of 1 (strongly disagree) to 5 (strongly agree).
Self-Regulation Questionnaire (SRQ) | Through study completion, an average of 14 weeks
  A self-report questionnaire that measures the ability to develop, implement, and flexibly maintain planned behavior. The extent to which the participant agrees with each statement is rated on a scale of 1 (strongly disagree) to 5 (strongly agree).
Self-Regulation Questionnaire (SRQ) | Study completion, an average of six to eight months
  A self-report questionnaire that measures the ability to develop, implement, and flexibly maintain planned behavior. The extent to which the participant agrees with each statement is rated on a scale of 1 (strongly disagree) to 5 (strongly agree).
Perceived Stress Scale (PSS) | Baseline
  A self-report questionnaire that measures the level of perceived stress for a participant. How often the participant experiences each event is rated on a scale of 0 (never) to 4 (very often).
Perceived Stress Scale (PSS) | Through study completion, an average of 14 weeks
  A self-report questionnaire that measures the level of perceived stress for a participant. How often the participant experiences each event is rated on a scale of 0 (never) to 4 (very often).
Perceived Stress Scale (PSS) | Study completion, an average of six to eight months
  A self-report questionnaire that measures the level of perceived stress for a participant. How often the participant experiences each event is rated on a scale of 0 (never) to 4 (very often).
Revised Helping Alliance Questionnaire (HAQ-II) | Through study completion, an average of 14 weeks
  A self-report questionnaire that measures the strength of the client therapist alliance. The extent to which the participant agrees with each statement is rated on a scale of 1 (strongly disagree) to 6 (strongly agree)
Moral Injury Events Scale (MIES) | Baseline
  A self-report survey that measures potentially morally injurious events. Each phrase is reacted on a Likert scale of 1 (Strongly Agree) to 6 (strongly disagree).
Moral Injury Events Scale (MIES) | Through study completion, an average of 14 weeks
  A self-report survey that measures potentially morally injurious events. Each phrase is reacted on a Likert scale of 1 (Strongly Agree) to 6 (strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Chandler Rhodes, PhD, Principal Investigator — WRNMMC
Locations (2):
- United States (2):
  - National Intrepid Center of Excellence, Bethesda, Maryland
  - ISC at Fort Belvoir, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No